CLINICAL TRIAL: NCT06212297
Title: A Clinical Trial to Evaluate the Safety and Efficacy of Subretinal Re-Administration of LX101 to the Contralateral Eye in Subjects With Biallelic RPE65 Mutation-associated Inherited Retinal Dystrophy
Brief Title: Fellow-eye Study (FE) of LX101 in Subjects With Inherited Retinal Dystrophy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNOSTELLAR-LX101-2
Record Dates: First submitted 2023-12-25; First posted 2024-01-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Inherited Retinal Dystrophy
Keywords: RPE65 Mutations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LX101 Subretinal Administration (Experimental)
  Interventions: Genetic: LX101

INTERVENTIONS:
Genetic: LX101 — Subretinal administration of LX101 to the contralateral, previously uninjected eye

SUMMARY:
Up to nine subjects who have participated in the earlier LX101 clinical study, and who meet all study eligibility criteria, will receive LX101 administration in the previously uninjected, contralateral eye to evaluate the safety of bilateral, sequential subretinal administration of LX101.

ELIGIBILITY:
Inclusion Criteria:

Prior subretinal administration of LX101 (unilateral)

≥ 6 years old Signed written informed consent

Exclusion Criteria:

Prior gene therapy except LX101 Active intraocular or periocular infections Lacking of sufficient surviving retinal cells Prior ocular surgery within six months Retinoid like compounds or precursors were taken within three months Complicating systemic diseases Clinically significant abnormal baseline laboratory values Using of any retinal toxic compounds

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events (AEs) and serious adverse events (SAEs) | 6 months
  Incidence of ocular and non-ocular AEs and SAEs following LX102 subretinal injection

SECONDARY OUTCOMES:
Full-field Light Sensitivity Threshold (FST) Test | 6 months、12 months
  Changes in light sensitivity from baseline, assessed by FST in log cd.s/m2
Visual Acuity | 6 months、12 months
  Changes in visual acuity from baseline, based on the ability to read letters using the Early Treatment Diabetic Retionpathy Study (ETDRS) chart
Mobility Test | 6 months、12 months
  Changes in functional vision from baseline, determined by mobility test score

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China